CLINICAL TRIAL: NCT04287738
Title: Care Ecosystem: Navigating Patients and Families Through Stages of Care, Extension Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Nebraska (Other); National Institute on Aging (NIA) (NIH); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01AG056715-01 (NIH); 1R01AG056715-01 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-02-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Lobar Degeneration; Memory Disorders
Keywords: Pragmatic Clinical Trial; Family Caregivers; Patient Care Management
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Lobar Degeneration; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigated Care (Experimental): Telephone-based collaborative dementia care navigation
  Interventions: Behavioral: Navigated Care
- Survey of Care (No Intervention): Control group that will receive usual care and undergo the same regular assessments as patients enrolled in Navigated Care

INTERVENTIONS:
Behavioral: Navigated Care — Telephone-based collaborative dementia care was delivered by a trained care team navigator, who provided education, support and care coordination with a team of dementia specialists (advanced practice nurse, social worker, and pharmacist). For more details, please see references below.
  Arms: Navigated Care

SUMMARY:
This is an extension trial of a prior trial (NCT02213458). Both persons with dementia (PWD) and their caregivers were enrolled as dyads. The purpose of this randomized clinical trial is to evaluate the benefits of a program that supports model care for PWD and their caregivers. Whereas the prior trial only delivered care and examined outcomes up to 12-months, this trial extends care and outcome measurement for 5 years or until death, and includes all dyads where the caregiver reported high caregiver burden (Zarit-12 greater than or equal to 17) at pre-randomization baseline for the original trial. Participants were recruited from California, Nebraska and Iowa. Participants determined to be eligible were consented and randomized into one of two groups. Two thirds of dyads were enrolled into Navigated Care that provided them with phone-based assistance in meeting important benchmarks in their care, for example completion of legal and financial planning and strategies for minimizing caregiver burden. One third of dyads were enrolled to a control group, entitled Survey of Care. Outcomes were unchanged from the original trial except for the addition of time to long term care placement and are detailed below.

ELIGIBILITY:
This study will enroll patients as well as their primary caregivers as research participants.

Inclusion criteria for patient participants:

* Patient has a diagnosis of dementia with a progressive course
* Patient has a primary caregiver (identified as having primary responsibility for patient) that is eligible for and agrees to join the study
* Patient is covered by Medicare or Medi-caid or is Medi-pending
* Patient is expected to live at least 3 months based on assessment by the referring provider, the patient's primary care provider, or medical record review
* Patient speaks English, Cantonese, or Spanish
* Patient lives in California or Nebraska or Iowa
* Patient is age 45 or older

Inclusion criteria for caregiver participants:

* Caregiver has primary responsibility for dementia patient that is eligible for and agrees to join the study
* Caregiver speaks English, Cantonese, or Spanish
* Caregiver is a legal adult
* Zarit-12 caregiver burden score greater than or equal to 17 at pre-randomization (baseline); this criteria is specific to this extension trial

Exclusion Criteria:

* Patient resides in a nursing home or skilled nursing facility at time of enrollment
* Participant is enrolled in a similar clinical trial that precludes their participation in the investigator's trial
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life - AD (Alzheimer's Disease) | From baseline to 60 months
  An established 13-item measure, with a 1-4 ordinal scale for each item, to obtain a rating of the patient's quality of life from the caregiver. Item scores are summed for a total score ranging from 13-52, with higher scores representing better quality of life

SECONDARY OUTCOMES:
Change in Health Care Utilization | From baseline to 60 months
  Health care utilization based upon caregiver survey to assess emergency department, hospitalization, and ambulance use rates. Measures number of times utilized, with higher scores indicating a worse outcome. To be confirmed using Medicare claims data.
Change in Zarit Burden Interview (short version). | From baseline to 60 months
  An established 12-item measure, with a 0-4 ordinal scale for each item, to measure caregiver burden. Item scores are summed for a total score ranging from 0-48, with higher scores representing higher levels of burden.
Change in Patient Health Questionnaire 9 (PhQ-9). | From baseline to 60 months
  An established 9-item measure administered to the caregiver. Higher scores represent more severe caregiver depression
Change in Caregiver Self-Efficacy: 1-5 ordinal scale | From baseline to 60 months
  A novel 4-item measure on a 1-5 ordinal scale to measure self-efficacy around dementia caregiving. Higher scores represent greater self-efficacy
Time to Long Term Care Placement | From date of baseline survey to immediately following long term care placement, assessed up to 60 months
  Number of days post randomization until nursing home or assisted living placement, excluding temporary stays

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Possin, Ph.D., Principal Investigator — University of California, San Francisco

REFERENCES:
- [Background] Guterman EL, Kiekhofer RE, Wood AJ, Allen IE, Kahn JG, Dulaney S, Merrilees JJ, Lee K, Chiong W, Bonasera SJ, Braley TL, Hunt LJ, Harrison KL, Miller BL, Possin KL. Care Ecosystem Collaborative Model and Health Care Costs in Medicare Beneficiaries With Dementia: A Secondary Analysis of a Randomized Clinical Trial. JAMA Intern Med. 2023 Nov 1;183(11):1222-1228. doi: 10.1001/jamainternmed.2023.4764. PMID 37721734
- [Background] Liu AK, Possin KL, Cook KM, Lynch S, Dulaney S, Merrilees JJ, Braley T, Kiekhofer RE, Bonasera SJ, Allen IE, Chiong W, Clark AM, Feuer J, Ewalt J, Guterman EL, Gearhart R, Miller BL, Lee KP. Effect of collaborative dementia care on potentially inappropriate medication use: Outcomes from the Care Ecosystem randomized clinical trial. Alzheimers Dement. 2023 May;19(5):1865-1875. doi: 10.1002/alz.12808. Epub 2022 Nov 4. PMID 36331050
- [Result] Possin KL, Merrilees JJ, Dulaney S, Bonasera SJ, Chiong W, Lee K, Hooper SM, Allen IE, Braley T, Bernstein A, Rosa TD, Harrison K, Begert-Hellings H, Kornak J, Kahn JG, Naasan G, Lanata S, Clark AM, Chodos A, Gearhart R, Ritchie C, Miller BL. Effect of Collaborative Dementia Care via Telephone and Internet on Quality of Life, Caregiver Well-being, and Health Care Use: The Care Ecosystem Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1658-1667. doi: 10.1001/jamainternmed.2019.4101. PMID 31566651
- [Result] Possin KL, Merrilees J, Bonasera SJ, Bernstein A, Chiong W, Lee K, Wilson L, Hooper SM, Dulaney S, Braley T, Laohavanich S, Feuer JE, Clark AM, Schaffer MW, Schenk AK, Heunis J, Ong P, Cook KM, Bowhay AD, Gearhart R, Chodos A, Naasan G, Bindman AB, Dohan D, Ritchie C, Miller BL. Development of an adaptive, personalized, and scalable dementia care program: Early findings from the Care Ecosystem. PLoS Med. 2017 Mar 21;14(3):e1002260. doi: 10.1371/journal.pmed.1002260. eCollection 2017 Mar. PMID 28323819
- [Result] Chen Y, Wilson L, Kornak J, Dudley RA, Merrilees J, Bonasera SJ, Byrne CM, Lee K, Chiong W, Miller BL, Possin KL. The costs of dementia subtypes to California Medicare fee-for-service, 2015. Alzheimers Dement. 2019 Jul;15(7):899-906. doi: 10.1016/j.jalz.2019.03.015. Epub 2019 Jun 4. PMID 31175026
- [Result] Merrilees JJ, Bernstein A, Dulaney S, Heunis J, Walker R, Rah E, Choi J, Gawlas K, Carroll S, Ong P, Feuer J, Braley T, Clark AM, Lee K, Chiong W, Bonasera SJ, Miller BL, Possin KL. The Care Ecosystem: Promoting self-efficacy among dementia family caregivers. Dementia (London). 2020 Aug;19(6):1955-1973. doi: 10.1177/1471301218814121. Epub 2018 Nov 29. PMID 30497302
- [Result] Guterman EL, Allen IE, Josephson SA, Merrilees JJ, Dulaney S, Chiong W, Lee K, Bonasera SJ, Miller BL, Possin KL. Association Between Caregiver Depression and Emergency Department Use Among Patients With Dementia. JAMA Neurol. 2019 Oct 1;76(10):1166-1173. doi: 10.1001/jamaneurol.2019.1820. PMID 31282955
- [Result] Bernstein A, Rogers KM, Possin KL, Steele NZR, Ritchie CS, Miller BL, Rankin KP. Primary Care Provider Attitudes and Practices Evaluating and Managing Patients with Neurocognitive Disorders. J Gen Intern Med. 2019 Sep;34(9):1691-1692. doi: 10.1007/s11606-019-05013-7. No abstract available. PMID 31044411
- [Result] Rosa TD, Possin KL, Bernstein A, Merrilees J, Dulaney S, Matuoka J, Lee KP, Chiong W, Bonasera SJ, Harrison KL, Kahn JG. Variations in Costs of a Collaborative Care Model for Dementia. J Am Geriatr Soc. 2019 Dec;67(12):2628-2633. doi: 10.1111/jgs.16076. Epub 2019 Jul 18. PMID 31317539
- [Result] Bernstein A, Harrison KL, Dulaney S, Merrilees J, Bowhay A, Heunis J, Choi J, Feuer JE, Clark AM, Chiong W, Lee K, Braley TL, Bonasera SJ, Ritchie CS, Dohan D, Miller BL, Possin KL. The Role of Care Navigators Working with People with Dementia and Their Caregivers. J Alzheimers Dis. 2019;71(1):45-55. doi: 10.3233/JAD-180957. PMID 31322558